CLINICAL TRIAL: NCT06162442
Title: Management of the Ocular Surface With Preservative-Free Lubricants in Patients With Dry Eye
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tecnoquimicas (Industry)
Responsible Party: Sponsor
Other Study IDs: CEI-001
Record Dates: First submitted 2023-09-27; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Propylene Glycol; Polyethylene Glycols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Preservative-free sterile ophthalmic solution, with 0.3% propylene glycol and 0.4% polyethylene glycol (400) — The procedures during the study consist of ophthalmological activities and attention to the participating subject with a diagnosis of DED and who starts using a specified ocular lubricant, free of preservatives. The ophthalmologist will notify the subject of the "wash out", which will consist of suspending the usual treatment medication for 7 days, to then start with the lubricant Glicolub Ultra®, with a dosage of 1 drop every 6 hours in both eyes. Self-assessment questionnaires will be delivered for their respective completion. An assessment will be made by the comprehensive ophthalmologist in all clinical tests for dry eye with a mild to moderate diagnosis, under compliance with the TOSF DEWS II criteria and study inclusion criteria.

SUMMARY:
Observational and prospective cohort study that seek to evaluate the epidemiological characteristics and changes in the ocular surface of patients diagnosed with dry eye disease who are treated with preservative-free lubricating drops.

DETAILED DESCRIPTION:
Question Research: What are the clinical and epidemiological characteristics of patients with dry eye treated with preservative-free lubricating drops at Clínica Sigma? JUSTIFICATION The true importance of dry eye lies in the great impact that it is having today throughout the world, both in the visual quality and in the life of those who suffer from it. Preservative-free lubricating drops are part of the treatment to alleviate the symptoms of DED and their management is becoming more frequent and improves for the patient due to the fewer reports of adverse events in their use. Currently, in Colombia there is little scientific evidence. In particular, at the regional level, there is no characterization of DED, which allows determining its causes for a timely diagnosis and adequate treatment of the patient. From the Sigma Clinic, knowing the epidemiological characterization of the population that consults for symptoms of mild to moderate dry eye, will allow establishing risk factors and evaluating the evolution of the disease with clinical staining tests and knowing the visual quality of the patient with the use of questionnaires. GENERAL OBJECTIVE: To describe the clinical and epidemiological characteristics of patients with mild to moderate dry eye treated with preservative-free lubricating drops at the Sigma Clinic. SPECIFIC OBJECTIVES: 1.Evaluate through OSDI and DEQ questionnaires the clinical evolution of patients diagnosed with mild to moderate dry eye treated with preservative-free lubricants from Clínica Sigma. 2. Assess the frequency and severity of symptoms with the SANDE questionnaire in patients with moderate to dry eye treated with preservative-free lubricants from Clínica Sigma. 3. Assess the quality of life with the NEI VFQ-25 questionnaire in patients with moderate to dry eye treated with preservative-free lubricants from Clínica Sigma.Prospective cohort study in patients with a previous diagnosis of mild dry eye and moderate dry eye, classified by DEWS II scale.

Those who wish to participate in the study will be informed at the first ophthalmological care of the need to withdraw the medication they were using for the usual treatment and start a wash-out for seven days. After seven days, the patient will start with the Glicolub Ultra® lubricant with a dosage of 1 drop every 6 hours in both eyes and the following three visits will be made by the study ophthalmologist in their 1st week, 3rd month and 6omes, with Glicolub Ultra® preservative-free lubricating drops. The information obtained will be recorded in the case report formats, initial CRF-1 and follow-up CRF-2, designed for this study and within the clinical history of the participating subject. During each of these services, the participating subjects will fill out the five self-assessment questionnaires, on the OSDI, SANDE, DEQ-5, NEI VFQ-25 scales and a similar tolerability scale (see annexes). The completion will be done online (after training the platform) or by print with an estimated duration of 30 to 40 minutes.

In turn, the participant agrees to return the Glicolub Ultra® vials used during the study to the main investigator. Which, will allow to determine the adherence to the treatment after its weighing and verification of use.

ELIGIBILITY:
Inclusion Criteria:

* Ability to sign informed consent.
* Any sex.
* Women of reproductive age should secure a method during the contraceptive study.
* Diagnosis of dry eye (mild, moderate) prior to the study in treatment with lubricants with preservatives.

Exclusion Criteria:

* Patients with any acquired or congenital anomaly or ocular malformation that prevents an adequate exploration of the ocular surface.
* Patients with a history of ocular surface surgery (cornea and conjunctiva).
* Patients being treated with medications that may compromise the state of the ocular surface: glaucoma, allergy, scarring diseases.
* Patients with allergy to fluorescein, lissamine green or tetracaine.
* Patients with lacrimal duct obstruction
* Severe dry eye
* Kidney failure
* Liver failure
* Pregnancy
* Breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with a previous diagnosis of mild to moderate dry eye from the dry eye unit of the Sigma Clinic, under the DEWS II criteria, being treated with lubricants with preservatives. Those who wish to participate in the study must have the drug with preservatives removed by washing or "wash out" for seven days and meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Age | At enrollment
  Years
Sex | At enrollment
  Genre: male, female, other
Medical history | At enrollment
  Presence or absence: Lupus, rheumatoid arthritis, scleroderma, Thyroid, none of above.
Occupation | At enrollment
  employee, independent, unemployed, other

SECONDARY OUTCOMES:
Scores Dry Eye Questionnaire: DEQ-5 | At enrollment, first week, third month and sixth month
  5 questions, scale 0 to 22, with higher score, representing greater disability
Scores Ocular Surface Disease Index Questionnaire: OSDI | At enrollment, first week, third month and sixth month
  Scale 0 to 100, with higher scores representing greater disability
National Eye Institute Visual Function Questionnaire de 25 ítems: NEI VFQ-25 | At enrollment, first week, third month and sixth month
  Scale 0 to 100, with 100 mm horizontal linear visual analog scale: 0 worse, to 100 is better
Scores Questionnaires: Symptom Assessment In Dry Eye (SANDE) | At enrollment, first week, third month and sixth month
  Horizontal linear visual analog scale. With more mm, more ocular symptoms
Scores Questionnaires DED: Questionaries: Visual Analog Scale (VAS) | At enrollment, first week, third month and sixth month
  Horizontal 0 to 100 mm linear visual analog scale. 0: worst and 100: better

OTHER OUTCOMES:
Ocular pressure | At enrollment, first week, third month and sixth month
  Measurement in mmHg. Normal between 10 - 20 mmHg; > 21 mmHg is anormal
Score ocular surface tests: TBUT | At enrollment, first week, third month and sixth month
  Tear breakup time: > 10 s, it is better, < 5 s, indicative of eye dry
Score ocular surface tests: Schirmer test | At enrollment, first week, third month and sixth month
  Assess tear production: distance of tear in filter paper. < 5 mm dry eye, > 10 mm normal

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Sigma, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No